CLINICAL TRIAL: NCT05350475
Title: Lymph Node Radiation Therapy with Integrated Boost to Prostate for High-risk Prostate Cancer a Randomized Phase 3 Trial Comparing Photons Vs. Protons
Brief Title: Protons Vs. Photons for High-risk Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Rigshospitalet, Denmark (Other); Odense University Hospital (Other); Aarhus University Hospital (Other); Aalborg University Hospital (Other); Sygehus Lillebaelt (Other); Herlev and Gentofte Hospital (Other); Naestved Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-10-72-290-21
Record Dates: First submitted 2022-03-16; First posted 2022-04-28 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2024-12

CONDITIONS: Prostate Cancer; Radiotherapy Side Effect
Keywords: Proton Therapy; High Risk; Intensity Modulated Radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms; Radiation Injuries | interventions — Proton Therapy

STUDY DESIGN:
Intervention Model Description: A randomized phase 3 study, randomizing 1:1 between photon vs. proton therapy for prostate cancer patients with high risk disease
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Proton therapy (Experimental): Radiation: Proton Therapy 78 Gray (Gy) in 39 fractions with 56 Gy to the Pelvic Lymph Nodes (LN), 5 days a week.
  Androgen Deprivation Therapy (ADT) for three years, starting 3 months before Proton Therapy.
  Interventions: Radiation: Proton therapy
- Photon Therapy (Active Comparator): Radiation: Photon Therapy 78 Gy in 39 fractions with 56 Gy to the pelvic LN, 5 days a week. ADT for three years, starting 3 months before Photon Therapy.
  Interventions: Radiation: Photon therapy

INTERVENTIONS:
Radiation: Proton therapy — Patients in the experimental arm will receive proton therapy within the same dose and fraction schedule as patients receiving photon therapy, which is standard treatment.
  Arms: Proton therapy
Radiation: Photon therapy — Patients in the photon arm will receive standard treatment with photon therapy.
  Arms: Photon Therapy

SUMMARY:
The purpose of this study is to assess late gastro-intestinal side-effects comparing proton therapy to photon therapy in high-risk prostate cancer patients receiving whole pelvic irradiation.

DETAILED DESCRIPTION:
Proton therapy (PT) is a radiation technique with possibility to spare normal pelvic organs: bladder, rectum and bowel for PC patients.

Most PC patients treated with PT receive PT to the prostate gland alone. With PT, we aim to examine PC patients in high risk with both lymph node and prostate treatment will experience less late side effects with PT compared to photon treatment.

The investigators propose a national open-labelled phase III randomized controlled trial (RCT) of proton therapy versus photon therapy of the prostate including the regional elective LN for localized/locally advanced prostate cancer patients combined with androgen deprivation therapy (ADT) aimed at 3 years. The investigators aim at reducing gastro-intestinal toxicity grad 2 more than 5 points, which is considered clinical significant, measured by mean Expanded Prostate Cancer Index Composite-26 (EPIC-26) bowel scores at 24 months and improve HRQOL. Secondary endpoints include morbidity, quality of life and survival data up to 10 years after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified localized/locally advanced prostate cancer T1-3bN0-1M0 (TNM 8th edition). A clinical T4 is allowed if it is because of invasion into the bladder neck.
* Adenocarcinoma (mixed histology allowed as long as the adenocarcinoma component comprise more than 50%)
* Indication for elective lymph node irradiation
* PSA < 100 ng/mL
* Age ≥18 years
* Performance status 0-1
* Life expectancy ≥ 10 years
* Able to understand and comply with the treatment protocol
* No evidence of inflammatory bowel disease Ability to adhere to procedures for study and follow-up
* Signed informed consent to participate in the study

Exclusion Criteria:

* No previous treatment for prostate cancer
* Hip-prostheses
* Other metal devices in the pelvic region (except fiducials)
* Previous major abdominal/rectal surgery
* Any other malignancy the last five years except for basal or squamous cell skin cancer
* Unable to understand patient information or comply with treatment and safety instructions
* Unable to read and understand patient information due to cognitive disabilities or language (Danish).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2037-03-01 (Estimated)

PRIMARY OUTCOMES:
Late gastrointestinal (GI) toxicity at year 2 compared to baseline using Expanded Prostate Cancer Index Composite-26 (EPIC-26) | 2 years
  Patient Reported Outcome The investigators aim at reducing gastro-intestinal toxicity grad 2 more than 5 points, which is considered clinically significant, measured by mean points, which is considered clinically significant.

SECONDARY OUTCOMES:
Late Genito-urinary (GU) and sexual toxicity ≥ 2 grade at year 2 and 5 compared to baseline (Common Terminology Criteria for Adverse Events (CTCAE) toxicity score (CTC_AE 5.0) | 5 years
  Physician Assessed Toxicity Number of Participants With Treatment-Related Adverse events as assessed by CTCAE v5.0
Late GU and sexual toxicity at year 2, 5 and 10 compared to baseline (EPIC-26) | 10 years
  Patient Reported Outcome using on-line questionnaire to assess this outcome measure
Late GI toxicity at year 5 compared to baseline (EPIC-26) | 5 years
  Patient Reported Outcome using on-line questionnaire to assess this outcome measure.aim at reducing gastro-intestinal toxicity grad 2 more than 5 points, which is considered clinically significant, measured by mean points, which is considered clinically significant
Acute GI at start, at the end of therapy and week 12 compared to baseline (EPIC-26) | 12 weeks
  EPIC-26
Acute GI at start, at the end of therapy and week 12 compared to baseline (CTC_AEv.5.0) | 12 weeks
  Physician Assessed Toxicity
Acute GU toxicity at start, at the end of therapy and week 12 compared to baseline (EPIC-26) | 12 weeks
  EPIC-26
Acute GU toxicity at start, at the end of therapy and week 12 compared to baseline (CTC_AE v.5.0) | 12 weeks
  Physician Assessed Toxicity
General health related quality of life (QoL) at year 2, 5 and 10 compared to baseline (EORTC QLQ-C30) | 10 years
  Patient Reported Outcome General health related quality of life (QoL) at year 2, 5 and 10 (EORTC QLQ-C30)
Biochemical progression free survival (BCR), (Phoenix criteria) | 10 years
  blood test
Non-biochemical progression free survival (by imaging) | 10 years
  Radiology assesments
Overall survival (OS) | 10 years
  Follow up

CONTACTS AND LOCATIONS:
Overall Officials: Stine Elleberg Petersen, MD, Ph.D, Principal Investigator — Danish Centre for Particle Therapy, Aarhus University Hospital
Locations (7):
- Denmark (7):
  - Dept. of Oncology, Rigshospitalet, Denmark, Copenhagen, Capital Region
  - Department of Oncology, Copenhagen University Hospital Herlev, Herlev, Capital Region
  - Department of Oncology, Aarhus University Hospital, Aarhus, Central Region
  - Dept. of Oncology, Aalborg University Hospital, Aalborg, Region North
  - Dept. of Oncology, Zealand University Hospital, Denmark, Næstved, Region Sjælland
  - Department of Oncology, Odense University Hospital, Odense, Region South
  - Department of Oncology, Vejle Hospital, Denmark, Vejle, Region South